CLINICAL TRIAL: NCT04619121
Title: Near-infrared Radiation-transcranial Photobiomodulation for Major Depressive Disorder: From Cellular, Animal Studies to a Sham-controlled Double-blind Randomized Clinical Trial
Brief Title: Near-infrared Radiation-transcranial Photobiomodulation for Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Ta-wei Guu, Attending physician, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMUH109-REC3-054
Record Dates: First submitted 2020-10-26; First posted 2020-11-06 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Major Depressive Disorder; Oxidative Stress
Keywords: near-infrared radiation-transcranial photobiomodulation; circadian rhythm; Inflammation; Brain energy metabolism
MeSH Terms: conditions — Depressive Disorder, Major; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with real NIR-tPBM on top of standing pharmacotherapy (Experimental): NIR t-PBM to the dorsolateral prefrontal cortex, bilaterally and simultaneously, from 20 minutes to 80 minutes a day, for 8 consecutive weeks.
  Interventions: Device: NIR-tPBM
- Sham device on top of standing pharmacotherapy (Sham Comparator): Sham device with neglectable energy to the dorsolateral prefrontal cortex, bilaterally and simultaneously, from 20 minutes to 80 minutes a day, for 8 consecutive weeks.
  Interventions: Device: Sham device

INTERVENTIONS:
Device: NIR-tPBM — The treatment will last for 8 weeks and be bilateral and applied to the frontal areas with one application site on the left side and one on the right side (left and right forehead centered on the frontal eminences and per EEG sites on F3 and F4). Energy is administered with a radiation wavelength of 830 nm. The duration of irradiation is from 20 minutes at each application site (the 2 sites are irradiated at the same time which is equivalent to 20 minutes of total time) to 40 minutes at each site, up to 2 times per day. The treatment will follow these specifications: PBM (IR) irradiance of 33.2 mW/cm2, each treatment window area is 28.7 cm2; PBM (IR) fluence of up to 60 Joules/cm2; energy delivered per session per device up to 1.72 kJ for a total of up to 3.44 kJ.
  Other Names: near-infrared transcranial photobiomodulation
  Arms: Treatment with real NIR-tPBM on top of standing pharmacotherapy
Device: Sham device — The sham device is completely identical in appearance, but only emits neglectable energy to the brain.
  Other Names: Sham
  Arms: Sham device on top of standing pharmacotherapy

SUMMARY:
This study was designed to be a 3 year, 3 phases project, and will explore the therapeutic effects from near-infrared transcranial photobiomodulation (NIR tPBM) in major depressive disordered human subjects, and it's biological mechanisms in cellular and animal model. However, due to shortage of funding under the pandemics, the project is now modified to start from its clinical part first, and will continue to its basic parts later when funding resources in place.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a leading cause of the overall global burden of disease in modern society, and has been estimated to move into the first place by 2030. Current antidepressants and psychotherapy had proved their efficacy, but are limited by the adverse effects and shortage of capable therapists worldwide. Accumulating evidence showed that hypometabolism of global and specific brain regions, inflammation, oxidative stress, suppression of neurogenesis and disturbed circadian rhythm all contribute to the pathophysiology of MDD.

Dr. Paolo Cassano, MD, PhD and his team from the Massachusetts General Hospital (MGH) of Harvard University recently demonstrated in both animal and human subjects that near-infrared radiation-transcranial photobiomodulation (NIR-tPBM) is a well-tolerated and effective treatment modality for MDD, and hypothesized NIR-tPBM may activate brain metabolism, be anti-inflammatory, reduce oxidative stress and promote neurogenesis. So far, the clinical studies are either open-labeled or only of small scale (n=21), and the real antidepressant mechanism of NIR-tPBM has not yet been fully understood. Adequately powered, well designed, double-blind randomized-control trials of larger scale is in pressing need.

In this 3-year study, we will collaborate with the team from Harvard University and MGH, to comprehensively evaluate from cellular mechanism, animal model, to clinical trials in human, the underlying mechanism of NIR-tPBM and the clinical strategy of NIR-tPBM. In the cellular study, we will culture and treat the human neuron-like cell lines with continuous NIR-PBM of different dosimetry and different duration, and compare the differences in cellular circadian rhythm, energy metabolism, and inflammation markers as well as the underlying gene expression. In the animal study, the mice under chronic stress environment will be treated with NIR-tPBM of different duration. We will compare the behavioral differences relevant to anxiety, depression and cognitive performance, as well as the differences in neurogenesis, neuroplasticity, energy metabolism, circadian rhythm, and inflammation markers of the mice and the gene expression of the biomarkers. In both cellular and animal studies, dose-response assessment will be applied. In the clinical human study, we will conduct a prospective, double-blind, randomized, sham-controlled trial, recruiting totally 80 MDD patients, age 18 to 75, and apply adjunctive NIR t-PBM to the dorsolateral prefrontal cortex, bilaterally and simultaneously, from 20 minutes and up to 80 minutes a day under the evaluation and recommendation of the clinicians, for 8 consecutive weeks. The change in depressive symptoms and circadian behaviors will be recorded in the 0, 2, 4, 8, 12 weeks and compared. The patient's peripheral blood-based biochemistry profile, inflammatory, oxidative stress, and circadian rhythm markers, as well as the gene expression of the relevant markers, will be collected in week 0, 8, and 12, and be compared.

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be included in the study only if they meet all of the following criteria:

  1. The subject should be between at least 18 years of age at screening, but has not had their 76th birthday at screening.
  2. Diagnosis of major depressive disorder (Based on Diagnostic Statistical Manual-IV or 5 ; diagnosis code: 296.22-296.23、296.32-296.33).
  3. HAM-D-17 ≥14 and ≤ 25
  4. Subject Informed Consent obtained in writing in compliance with local regulations prior to enrollment into this study.
  5. The subject (and caregiver, if applicable) is willing to participate in this study for at least 12 weeks.
  6. Subjects may only be taking one (1) antidepressant, and will need to be on a stable dose for at least four weeks prior to enrollment.

Exclusion Criteria:

* Subjects will be excluded from the study for any of the following reasons:

  1. The subject is pregnant or lactating.
  2. The subject failed two or more FDA-approved antidepressants during current episode.
  3. Structured psychotherapy focused on treating the subject's depression is exclusionary unless the subject has had at least 8 weeks of treatment prior to the screening visit.
  4. Substance used disorder in the past 6 months.
  5. Psychotic disorder or psychotic episode (current psychotic episode per assessment).
  6. Bipolar affective disorder (per assessment).
  7. Unstable or active medical illness.
  8. Active suicidal or homicidal ideation.
  9. The subject has a significant skin condition (i.e., hemangioma, scleroderma, psoriasis, rash, open wound or tattoo) on the subject's scalp that is found to be directly below any of the procedure sites.
  10. The subject has an implant of any kind in the head (e.g. stent, clipped aneurysm, embolized AVM, implantable shunt - Hakim valve).
  11. Any use of light-activated drugs (photodynamic therapy) within 14 days prior to study enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms (subjective) | Measured biweekly up to 12 weeks.
  Measured with Beck Depression Rating scale, value from 0 to 63, with higher scores indicating greater severity of depression.
Change in depressive symptoms (objective) | Measured biweekly until trial completed, up to 12 weeks.
  Measured with Hamilton Depression rating scale (21-items), value from 0 to 66, with higher scores indicating greater severity of depression.

SECONDARY OUTCOMES:
Change in circadian rhythm | Measured biweekly up to 12 weeks.
  Measured with Munich ChronoType Questionnaire (MCTQ), value of 16 to 86. It offers methods to make up for sleep log, and measures the behavioral change around the clock.
Change in sleep quality | Measured twice a week up to 12 weeks.
  Measured with Pittsburgh Sleep Quality Index,value of 0 to 21, provides a subjective measure of sleep quality and patterns. The higher the score, the worse the quality.

CONTACTS AND LOCATIONS:
Overall Officials: Ta-Wei Guu, MD, Principal Investigator — China Medical University, Taiwan
Locations (1):
- China Medical University Beigang Hospital, Beigang, Yunlin County, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Will be discussed internally after trial completed.

REFERENCES:
- [Background] Caldieraro MA, Cassano P. Transcranial and systemic photobiomodulation for major depressive disorder: A systematic review of efficacy, tolerability and biological mechanisms. J Affect Disord. 2019 Jan 15;243:262-273. doi: 10.1016/j.jad.2018.09.048. Epub 2018 Sep 17. PMID 30248638
- [Background] Salehpour F, Cassano P, Rouhi N, Hamblin MR, De Taboada L, Farajdokht F, Mahmoudi J. Penetration Profiles of Visible and Near-Infrared Lasers and Light-Emitting Diode Light Through the Head Tissues in Animal and Human Species: A Review of Literature. Photobiomodul Photomed Laser Surg. 2019 Oct;37(10):581-595. doi: 10.1089/photob.2019.4676. Epub 2019 Sep 25. PMID 31553265
- [Background] Cassano P, Caldieraro MA, Norton R, Mischoulon D, Trinh NH, Nyer M, Dording C, Hamblin MR, Campbell B, Iosifescu DV. Reported Side Effects, Weight and Blood Pressure, After Repeated Sessions of Transcranial Photobiomodulation. Photobiomodul Photomed Laser Surg. 2019 Oct;37(10):651-656. doi: 10.1089/photob.2019.4678. PMID 31647774
- [Background] Cassano P. Photomedicine and Pharmaceuticals: A Brain New Deal. Photobiomodul Photomed Laser Surg. 2019 Oct;37(10):575-576. doi: 10.1089/photob.2019.4733. Epub 2019 Sep 24. No abstract available. PMID 31549918
- [Derived] Guu TW, Cassano P, Li WJ, Tseng YH, Ho WY, Lin YT, Lin SY, Chang JP, Mischoulon D, Su KP. Wearable, self-administered transcranial photobiomodulation for major depressive disorder and sleep: A randomized, double blind, sham-controlled trial. J Affect Disord. 2025 Mar 1;372:635-642. doi: 10.1016/j.jad.2024.12.065. Epub 2024 Dec 18. PMID 39706483